CLINICAL TRIAL: NCT05401968
Title: Osteoporosis Patient Education in Danish Municipalities: an Evaluation of Existing Programs and Recommendations for Further Practice
Brief Title: Osteoporosis Patient Education in Denmark
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: National Research Center for Bone Health (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19/33410
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Osteoporosis
Keywords: Patient education
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: The municipalities recruit and include citizens in osteoporosis patient education. We have already received information on participants from 2016 until 2020, and thereafter we will create a matched control group, who have not participated in osteoporosis patient education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Osteoporosis patients who have participated in patient education
  Interventions: Behavioral: Osteoporosis patient education
- Control group (No Intervention): Osteoporosis patients who have not participated in patient education

INTERVENTIONS:
Behavioral: Osteoporosis patient education — During osteoporosis patient education the participants get knowledge about e.g. osteoporosis, medication, and diet, and they participate in physical exercises. Though, differences between municipalities exist. The participants meet in groups and face-to-face.
  Arms: Intervention group

SUMMARY:
In an effect evaluation the investigators will examine the effects of participating in osteoporosis patient education. An intervention group who have already participated in patient education will be compared to a matched control group who have not participated. Effects on quality of life, fractures, daily functional capacity, self-efficacy, psychological wellbeing, physical function, balance, falls, pain management, and adherence will be examined.

DETAILED DESCRIPTION:
In this quasi-experimental study the investigators will conduct an effect evaluation that compares an intervention group of osteoporosis patients who have participated in patient education in a municipality with a control group who have not participated.

The intervention group consists of citizens who have already participated in osteoporosis patient education from 2016 until 2020. The investigators have received information on the intervention group from the municipalities who store data on previous participants.

The control group will be extracted via the Danish Health Data Authority and consists of citizens who have not participated in osteoporosis patient education. For each individual in the intervention group one control will be matched regarding gender, age, diagnosis, time of diagnose, and type of fracture before the index date (i.e. the date the individual in the intervention group started on patient education).

The aim of the effect evaluation is to examine the effects of osteoporosis patient education on quality of life, fractures, daily functional capacity, self-efficacy, psychological wellbeing, physical function, balance, falls, pain management, and adherence.

Data is generated from a register extraction and a questionnaire-based survey. The questionnaire will include information on quality of life, daily functional capacity, self-efficacy, psychological wellbeing, physical function, balance, falls, and pain management. As far as possible validated questionnaires will be included to measure these outcomes. The register extraction will be made by the Danish Health Data Authority and include information on fractures and adherence.

All analyses are performed using Stata. In the analyses the investigators will compare the intervention group and the control group with regard to all outcomes. The covariates are selected on the basis of Directed Acyclic Graphs (DAG) and they include e.g. socioeconomic status, cohabitee status, and co-morbidity. The analysis will be completed on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* To participate in osteoporosis patient education in municipalities the participants should have osteoporosis or in few cases osteopenia.

Exclusion Criteria:

* None though this may vary across municipalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3132 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Differences in quality of life between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with the 12-item Short-Form Health Survey of the Medical Outcomes Study (SF-12)
Differences in clinical diagnosis of fracture between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Including hip, vertebral, forearm, and upper arm fractures registered in the National Patient Register

SECONDARY OUTCOMES:
Differences in daily functional capacity between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with questions from the European Health Interview Survey
Differences in self-efficacy between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with the questionnaire Self-Efficacy for Managing Chronic Disease 6-Item Scale (SES6G)
Differences in psychological well-being between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with the questionnaire Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS)
Differences in physical function between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with questions from The Danish National Health Survey
Differences in balance between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with self-constructed, validated questions regarding problems with balance and balance confidence
Differences in falls between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with self-constructed, validated questions regarding number of falls and concerns about falling
Differences in pain management between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Measured with the Pain Self-Efficacy Questionnaire (PSEQ)
Differences in adherence by Medication Possession Ratio (MPR) between intervention and control group | At follow-up (1 to 6 years after the index date i.e. the date the individual in the intervention group started on patient education)
  Including adherence to alendronate and ibandronate attained from the Danish National Prescription Registry

CONTACTS AND LOCATIONS:
Overall Officials: Holmberg, Principal Investigator — University of Southern Denmark; Andersen, Principal Investigator — University of Southern Denmark; Hitz, Principal Investigator — National Research Center for Bone Health
Locations (1):
- National Institute of Public Health, University of Southern Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
If possible, we will store data at The Danish National Archives. We will apply for storing at a later date.